CLINICAL TRIAL: NCT06578663
Title: Electrical Dry Needling Versus Iontophoresis in Treating Chronic Unilateral Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Ahmed Fayez Zehiry, lecturer assistant, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Horus_Phd_2024
Record Dates: First submitted 2024-05-16; First posted 2024-08-29 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail, repeated measured; pre and post-test experimental design will be conducted
Who Masked: Participant
Masking Description: The sample will be randomly divided into three groups: A, B, and C. Group A: The control group (n=20) Group B: The study group (n=20) will receive conventional physical therapy plus electrical dry needling.
  Group C: The study group (n=20) will receive conventional physical therapy plus glucosamine sulfate iontophoresis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional program (Sham Comparator): will receive conventional physical therapy, including transcutaneous electrical nerve stimulation (TENS) and an exercise therapy program (stretching exercises, both hip and knee strengthening, balance, and stability exercise)
  Interventions: Other: conventional physical therapy
- dry needling and conventional program (Experimental): will receive conventional physical therapy, plus electrical dry needling.
  Interventions: Other: conventional physical therapy; Other: Electrical Dry Needling
- Glucosamine sulfate iontophoresis and conventional program (Experimental): will receive conventional physical therapy, plus Glucosamine sulfate iontophoresis.
  Interventions: Other: conventional physical therapy; Other: Glucosamine sulfate iontophoresis

INTERVENTIONS:
Other: conventional physical therapy — including transcutaneous electrical nerve stimulation (TENS) and an exercise therapy program (stretching exercises, both hip and knee strengthening, balance, and stability exercise)
Other: Electrical Dry Needling — In electrical dry needling, needle electrodes are used to deliver an electric current to the taut muscle band or the pain-generating trigger point. Low-frequency currents are thought to improve the physiological effects of the therapy by using electrical stimulation to enhance certain physiological reactions and achieve a speedier analgesic and anesthetic effect than that obtained with standard dry needling.
  Arms: dry needling and conventional program
Other: Glucosamine sulfate iontophoresis — Galvanic current mode will be used to deliver the cream through the skin. One gram of GS will be placed on positive electrode (being positively charged using Trans-arthral electrode placement technique) for administration of Iontophoresis [40mA-min (2mA x 20minutes)].
  Arms: Glucosamine sulfate iontophoresis and conventional program

SUMMARY:
The goal of this clinical trial is to compare the effects of electrical dry needling versus glucosamine sulfate iontophoresis on pain intensity level, functional ability, and knee range of motion in chronic unilateral knee osteoarthritis patients.

DETAILED DESCRIPTION:
Knee Osteoarthritis (OA) is a chronic disease affecting 240 million people worldwide, with a higher prevalence in older adults. The disease leads to knee deformity, laxity, and ligament instability. Dry needling, a new treatment modality, uses needle electrodes to deliver an electric current to the pain-generating trigger point, improving the physiological effects and analgesic and anesthetic effects. Iontophoresis, a safer method of drug therapy, has shown to be more effective in pain reduction in knee osteoarthritic patients. The study aims to investigate the effect of electrical dry needling versus glucosamine sulfate iontophoresis on pain intensity level, knee function, and range of motion (ROM) in chronic knee OA patients. This approach aims to maximize drug bioavailability, optimize therapeutic efficacy, and minimize side effects.

ELIGIBILITY:
Inclusion Criteria:

1. The patient will be selected from the outpatient clinic of physical therapy at Horus University, New Damietta, Egypt, diagnosed with a Kellgren/Lawrence grade 2,3 radiological severity of knee osteoarthritis (OA). and referred by an orthopedist.
2. Age will range from 40 to 60 years.
3. Body mass index will range from 25 to 29.9 kg/m2.
4. Duration of knee pain not less than 3 months prior to study .

Exclusion Criteria:

1. Patients with history of cardiac disorder with pacemaker.
2. Knee surgery.
3. Diabetes and nutritional disorder.
4. Neuromuscular and other musculoskeletal diseases.
5. Any red flags to dry needling, or conventional therapy.
6. Had received physical therapy, acupuncture, massage therapy, chiropractic, or intra-articular injections for the painful knee in the last 3 months.
7. Presented with positive neurological signs.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity level measurement | at baseline and after 6 weeks
  The visual analog scale (VAS) is a pain rating scale .A 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)
Functional ability measurement | at baseline and after 6 weeks
  Knee Injury and Osteoarthritis Outcome (KOOS) Score.A 0-100 scale, with zero express extreme knee problems and 100 for no knee problems, as common in orthopedic scales.
Knee ROM measurement | at baseline and after 6 weeks
  A digital goniometer will be used to measure active knee ROM. The subject will be supine, flexing and extending their knee to the maximum. Bony landmarks will be identified for standardization and repeatability. The goniometer will be positioned over the lateral epicondyle of the femur, with the greater trochanter for reference. Measurements will be made three times, and the average value will be analyzed. Knee ROM measurements in patients with knee OA show high reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Horus university, Damietta, Egypt